CLINICAL TRIAL: NCT05129852
Title: The Effect Of Reiki And Massage With Sage Oil On Pain In Young Girls With Primary Dysmenorrhea
Brief Title: The Effect Of Reiki And Massage With Sage Oil On Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, NAZİFE BAKIR, Assistant Professor,, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAKU-BSYO-NB-01
Record Dates: First submitted 2021-10-29; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Primary Dysmenorrhea
Keywords: midwifery, nurse, alternative therapies

STUDY DESIGN:
Intervention Model Description: Three groups with alternative therapy is a randomized controlled trial
Who Masked: Participant
Masking Description: The researchers massaged the abdomen with sage oil for 30 minutes, and 30 minutes after the massage, VAS evaluation and blood pressure, body temperature, and pulse rate measurements were performed again.
  VAS pain scores were also evaluated in the Reiki group (30 participants) when the pain started. The participants experienced pain on the first 3 days of their menstruation. Their blood pressure, body temperature, and pulse rate were also measured. Reiki was applied by a researcher with a Reiki certificate. Thirty minutes after the Reiki application, VAS evaluation and blood pressure, body temperature, and pulse rate measurements were repeated. This application was repeated for two menstrual periods.
  Similarly, in the control group (30 participants), VAS pain scores were evaluated when the pain started on the first three days of their menstruation, and their blood pressure, body temperature, and pulse rate were measured. No application was performed; they were only asked to rest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sage oil group (Active Comparator): The participants in the sage oil massage group (30 participants in total) had pain in the first 3 days of their menstrual cycle; when the pain started, pain levels were scored by the participants using visual analog scale (VAS). In addition, their blood pressure, body temperature, and pulse rate were measured. The researchers massaged the abdomen with sage oil for 30 minutes, and 30 minutes after the massage, VAS evaluation and blood pressure, body temperature, and pulse rate measurements were performed again. This application was repeated for two menstrual periods.
  Interventions: Other: Sage oil group
- Reiki group (Active Comparator): visual analog scale (VAS) pain scores were also evaluated in the Reiki group (30 participants) when the pain started. The participants experienced pain on the first 3 days of their menstruation. Their blood pressure, body temperature, and pulse rate were also measured. Reiki was applied by a researcher with a Reiki certificate. Thirty minutes after the Reiki application, VAS evaluation and blood pressure, body temperature, and pulse rate measurements were repeated. This application was repeated for two menstrual periods.
  Interventions: Behavioral: Reiki group
- control group (No Intervention): Similarly, in the control group (30 participants),visual analog scale (VAS) pain scores were evaluated when the pain started on the first three days of their menstruation, and their blood pressure, body temperature, and pulse rate were measured. No application was performed; they were only asked to rest. VAS evaluation and blood pressure, body temperature, and pulse rate measurements were performed again after 30 minutes. These measurements were repeated for two menstrual cycles.

INTERVENTIONS:
Other: Sage oil group — Sometimes called muscatel. Made by steam or water distillation of Salvia sclarea flowering tops and foliage. Yields range from 0.7 to 1.5%. A pale yellow to yellow liquid with a herbaceous odor and a winelike bouquet. Produced in large quantities in France, Russia and Morocco. The oil contains linalyl acetate, linalool and other terpene alcohols (sclareol), as well as their acetates.
  Arms: sage oil group
Behavioral: Reiki group — Within complementary and integrative health practices, Reiki is an ancient practice of Japanese origin widely used worldwide. Through the touch or approximation of the hands, an enabled therapist applies this technique to eliminate toxins, to balance the organism, and to favor the full functioning of the organism, to reestablish the flow of vital energy. Reiki as bioenergy therapy works with the energy that leads the human body to a calmer state that is linked to health and cure. Reiki therapists conduct the curing energy that enters the top of the head and leaves through the hands.
  Arms: Reiki group

SUMMARY:
This study was a randomized controlled trial. It included young girls with primary dysmenorrhea in a district located in the south of Turkey and was conducted between March 01, 2021 and June 30, 2021. The sample size of this research was decided by performing a power analysis in the power statistical program. Considering the parameters of the groups, the effect size was calculated to be 0.5003604. Since α was found to be 0.05 and power (1 - β) was 0.95, a total number of 66 participants were distributed into three equal groups (sage oil massage: 22, Reiki: 22, control: 22). Considering the possibility of case losses, 30 participants were included in each group; finally, a total of 90 people were included in the study. For data collection, a questionnaire regarding sociodemographic characteristics and the visual analog scale (VAS) were used. Reiki and massage with sage oil were applied for 30 minutes, and no application was performed on the control group.

ELIGIBILITY:
Inclusion Criteria:

Being female Not married

Exclusion Criteria:

Psychiatric problem Communication barrier Those who refuse to work

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 90 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Individual Introductory Information Form | 2 months
  Form, information regarding sociodemographic characteristics of the participants was collected.
VAS pain scores | 2 months
  Pain levels were scored by the participants using VAS
Body Mass Index | 2 months
  Body mass index was calculated by measuring the height and weight of the participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Nazife Bakir, Burdur, Bucak, Turkey (Türkiye)